CLINICAL TRIAL: NCT00210197
Title: Plasma Coagulation Parameters and Hypercoagulability After Breast Cancer Surgery
Brief Title: Hypercoagulability After Breast Cancer Surgery
Acronym: EHC
Status: Completed | Type: Observational
Sponsor: Institut Bergonié (Other)
Other Study IDs: IB2005-06; EHC
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2007-10

CONDITIONS: Breast Cancer; Blood Coagulation Disorders
Keywords: Hypercoagulability; Plasma coagulation parameters; Breast cancer
MeSH Terms: conditions — Breast Neoplasms; Blood Coagulation Disorders; Thrombophilia | interventions — Lead

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: Blood collection (pre and postoperative): plasma coagulation parameters

SUMMARY:
The risk of deep venous thrombosis after radical breast surgery is known. The objective of this study is to explore hypercoagulability after radical breast cancer surgery by studying several factors for haemostasis before, during and after surgery. Ultrasound Doppler examination is realised between 24 and 72 hours post-operatively. Hypercoagulability is defined by a significant increasing level of thrombin-antithrombin, D-dimer and the endogen thrombin potential.

ELIGIBILITY:
Inclusion criteria:

* Breast cancer
* mastectomy

Exclusion criteria:

* thrombophilia
* anticoagulant treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast Cancer
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2005-01; Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Youssef KABBANI, MD, Principal Investigator — Institut Bergonié
Locations (1):
- Institut Bergonié - Centre Régional de Luttre Contre le Cancer de Bordeaux et du Sud Ouest, Bordeaux, France